CLINICAL TRIAL: NCT01191840
Title: A Multi-Center, Randomized, Open-Label, Comparative Study to Assess the Safety and Efficacy of a Treatment Algorithm to Reduce the Use of Vancomycin in Adult Patients With Blood Stream Infections Due to Staphylococci
Brief Title: Treatment Algorithm to Reduce the Use of Vancomycin in Adults With Blood Stream Infection
Acronym: Bacteremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025497; DMID Protocol Number: 09-0080 (Other Grant/Funding Number: HHSN272200900023C)
Record Dates: First submitted 2010-08-28; First posted 2010-08-31 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Bacteremia
Keywords: staphylococci
MeSH Terms: conditions — Bacteremia | interventions — Vancomycin; Nafcillin; Oxacillin; Cloxacillin; Daptomycin; Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Algorithm-determined therapy (Experimental)
  Interventions: Drug: Vancomycin
- Standard of Care (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Duration
  Other Names: Nafcillin; Oxacillin; Cloxacillin; Daptomycin; Cefazolin
  Arms: Algorithm-determined therapy
Drug: Vancomycin — Duration
  Other Names: Nafcillin; Oxacillin; Cloxacillin; Daptomycin; Cefazolin
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to accurately determine the length of appropriate drug treatment for staphylococcal blood stream infection. The study seeks to address important information about the management of staphylococcal blood stream infections.

DETAILED DESCRIPTION:
To demonstrate that the clinical efficacy of algorithm-based therapy of patients with staphylococcal blood stream infection is noninferior to current standard of care.

PP (per protocol) population: randomized patients EXCLUDING those that: Received a PENS antibiotic -Did not undergo removal of intravascular catheter suspected to be infected. Note that patients with simple CoNS bacteremia may retain the catheter; all other patients should have their catheter(s) removed. -Had blood stream infection with a vancomycin-resistant staphylococcus; or a staphylococcus resistant to protocol-identified alternative drugs if these were used -Discontinued study medication prematurely for reasons other than clinical failure -Did not undergo final TOC assessment -Did not comply with all Patient Inclusion Criteria -Violated any Patient Exclusion Criteria

* Died within 3 days of randomization
* Were classified as non-evaluable

PPE Population: Patients from the PP population who did not have complicated staphylococcal infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent. The patient's legally authorized representative (LAR) can provide a signed informed consent for the patient if allowed by local Institutional Review Board/Ethics Committee (IRB/EC) policy.
2. Is ≥ 18 yrs of age.
3. If the subject has an intravenous catheter in place then the subject and his/her primary health care provider must agree to have the catheter removed within 5 days of the initial blood culture draw with the exception of those subjects who meet criteria for simple CoNS bacteremia as defined in Table 1. The catheter may be retained in those subjects with simple CoNS bacteremia.
4. Has blood stream infection defined as at least one blood culture positive for S. aureus or CoNS. In most cases, vancomycin(or other study drug alternative) will have been started prior to randomization. Enrollment windows depend on speciation and clinical classification as follows:

   1. identification of CoNS and classification as simple per Table 1-must be randomized within 3 calendar days of the start of treatment effective for the baseline infecting pathogen
   2. identification of CoNS and classification as uncomplicated per Table 1 must be randomized within 4 calendar days of the start of treatment effective for the baseline infecting pathogen
   3. identification of S. aureus - must be randomized within 12 calendar days of the start of treatment effective for the baseline infecting pathogen
5. This criterion has been removed
6. Women of child bearing potential must have a negative urine and/or serum pregnancy test.
7. All patients of reproductive potential must be abstinent or agree to use double-barrier contraception while receiving study (algorithm based or Standard of Care) therapy.

Exclusion Criteria:

1. Has known or suspected new complicated staphylococcal infection at the time of enrollment.
2. Weigh ≥ 200 kg.
3. Has non-removable intravascular foreign material at the time a positive blood culture was drawn (e.g., intracardiac pacemaker or cardioverter/defibrillator wires, hemodialysis access grafts, cardiac prosthetic valve, valvular support ring). Exception: coronary stents, inferior vena cava (IVC) filters in place > 6 weeks, patients with pacemakers whose baseline infecting pathogen is a CoNS, vascular stents in place for > 6 weeks, non-hemodialysis grafts in place >90 days and hemodialysis grafts not used within past 12 months and not previously infected are eligible for randomization. Arthroplasties and other extravascular devices, e.g. synthetic hernia repair mesh, and non-arthroplasty orthopedic prostheses including pins or plates, are acceptable as long as there are no signs or symptoms of foreign material-related infection at the time of randomization.
4. This criterion has been removed
5. Has a moribund clinical condition such that there is a high likelihood of death or cardiac surgery during the next three days.
6. Has shock or hypotension (supine systolic blood pressure < 80 mmHg) or oliguria (urine output < 20 mL/h) unresponsive to fluids or pressors within four hours.
7. Has received an investigational antibacterial agent with anti-staphylococcal activity within 30 days prior to randomization.
8. Has a documented history of significant allergy or intolerance to all protocol-approved antibiotics anticipated to be effective for their infection.
9. Has an infecting pathogen with confirmed reduced susceptibility to vancomycin (Minimum Inhibitory Concentrations (MIC) > 2 µg/mL) if known. Note: If reduced susceptibility to vancomycin is discovered after enrollment, the patient will be treated with daptomycin (if pathogen is susceptible). Patient will remain in study as appropriate and be evaluated in the Intent to Treat (ITT) analysis, but will be excluded from Protocol Population (PP) analyses.
10. For S. Aureus patients, is severely neutropenic (absolute neutrophil count < 0.100x103/mm3) or is anticipated to develop severe neutropenia (absolute neutrophil count < 0.100x103/ mm3) during the study treatment period due to prior or planned chemotherapy. CoNS patients with neutropenia are eligible to be enrolled.
11. This criterion has been removed
12. Has previously known Human Immunodeficiency Virus (HIV) infection with a nadir CD4+ count of <100 cells/mm3 within the past 12 months
13. Is considered unlikely to comply with study procedures or to return for scheduled post-treatment evaluations.
14. Is pregnant or trying to get pregnant, nursing, or lactating.
15. Has known or suspected septic arthritis, osteomyelitis, pneumonia or other metastatic focus of infection. CoNS patients with pneumonia and not being treated or anticipated to start treatment with antibiotics effective for the baseline infecting pathogen can be included
16. Has polymicrobial blood stream infection including at least one non-staphylococcal species, except AFTER consultation with the Clinical Medical Monitor at DCRI. Note that it is possible that a subject may not have a known polymicrobial bloodstream infection at the time of randomization, but additional pathogen(s) can subsequently be isolated from the initial blood culture. These patients will be eligible to remain in the trial. Please also note that patients with S. aureus plus CoNS will follow the treatment pathway for S. aureus.
17. This criterion has been removed.
18. Is hemodialysis dependent or has end stage renal disease (Creatinine Clearance (CrCl) < 30 cc/min).
19. Developed Staphylococcus aureus blood stream infection within 72 hours of percutaneous coronary revascularization
20. Received of any of the following antibiotics for 7 or more of the 10 calendar days immediately preceding the calendar day that the initial positive blood culture was drawn:

    1. If methicillin susceptibility of the isolate is unknown at the time of enrollment: vancomycin; daptomycin; telavancin; tigecycline; linezolid (in either oral or IV administration); quinupristin/dalfopristin; piperacillin/tazobactam; penicillin; nafcillin; oxacillin; cloxacillin; cefazolin, ceftriaxone, ceftaroline, dalbavancin, oritavancin, tedizolid, and levofloxacin or equivalent fluoroquinolone (in either oral or IV administration) Note: ciprofloxacin is not an exclusion criteria.
    2. If the staphylococcal isolate is known to be methicillin resistant: vancomycin; daptomycin; telavancin; tigecycline; linezolid (in either oral or IV administration), quinupristin/dalfopristin, dalbavancin, oritavancin, tedizolid, and ceftaroline.

    Note: patients who have developed bacteremia after at least 7 days of prophylaxis with oral antibiotics have by definition failed prophylaxis and the oral antibiotic can be deemed non-effective for the index bacteremia. Oral antibiotics that have failed as prophylaxis in this manner will not be considered exclusionary or count towards the number of antibiotic days but must be stopped upon randomization
21. Has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2011-02; Primary Completion 2017-03-04 (Actual); Study Completion 2017-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vance Fowler, MD, Principal Investigator — Duke University
Locations (15):
- United States (14):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Mass, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albert Einstein College of Medicine, The Bronx, New York
  - Carolina Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at ECU, Greenville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - UT MD Anderson Cancer Center, Houston, Texas
- Fundacio Clinic Privada per a la Recera, Barcelona, Spain

REFERENCES:
- [Derived] Holland TL, Raad I, Boucher HW, Anderson DJ, Cosgrove SE, Aycock PS, Baddley JW, Chaftari AM, Chow SC, Chu VH, Carugati M, Cook P, Corey GR, Crowley AL, Daly J, Gu J, Hachem R, Horton J, Jenkins TC, Levine D, Miro JM, Pericas JM, Riska P, Rubin Z, Rupp ME, Schrank J Jr, Sims M, Wray D, Zervos M, Fowler VG Jr; Staphylococcal Bacteremia Investigators. Effect of Algorithm-Based Therapy vs Usual Care on Clinical Success and Serious Adverse Events in Patients with Staphylococcal Bacteremia: A Randomized Clinical Trial. JAMA. 2018 Sep 25;320(12):1249-1258. doi: 10.1001/jama.2018.13155. PMID 30264119

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Drugs used to treat the bacteremia and the duration of treatment will be determined by the patient's primary medical provider.
- Algorithm-determined Therapy: Patients will be treated with Vancomycin or protocol-approved alternate antibiotic for 14 (-/+2) days for uncomplicated S. aureus, or 28-42 (-/+2) days if complicated S. aureus develops within the treatment period after randomization. Simple CoNS will be treated for 0 - 3 (+1) days, uncomplicated CoNS will be treated for 5 (-/+1) days, or 7-28 (-/+2) days if complicated CoNS develops within the treatment period after randomization.
Period: Overall Study
Arm/Group | Standard of Care | Algorithm-determined Therapy
Started | 254 | 255
Completed | 240 | 240
Not Completed | 14 | 15
Not completed — withdrew consent | 2 | 1
Not completed — Subject discontinued treatment | 1 | 2
Not completed — Lost to Follow-up | 4 | 6
Not completed — Non Staph Infection | 4 | 3
Not completed — ineligible at enrollment | 1 | 0
Not completed — IRB approval lapse | 0 | 2
Not completed — lab error speciation - non Staph infecti | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Algorithm-determined Therapy | Total
Number analyzed (Participants) | 254 | 255 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (17.1) | 55.8 (16.5) | 56.6 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 109 | 226
  Male | 137 | 146 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 44
  Not Hispanic or Latino | 231 | 234 | 465
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 1 | 2
  Race: Asian | 4 | 2 | 6
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: Black or African American | 60 | 63 | 123
  Race: White | 174 | 175 | 349
  Race: More than one race | 2 | 4 | 6
  Race: Other | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate
Description: To compare the cure rate at Test of Cure evaluation, between the proposed treatment algorithm and the standard of care therapy.
Time Frame: Test of cure 2 (up to approximately 42 days)
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Algorithm-determined Therapy
Number analyzed (Participants) | 254 | 255
Participants | 207 | 209

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of Participants that reported a Serious Adverse Event
Time Frame: Test of cure 2 (up to approximately 42 days)
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Algorithm-determined Therapy
Number analyzed (Participants) | 254 | 255
Participants | 72 | 83

3. Primary Outcome: Number of Participants With Adverse Events Leading to Study Drug Withdrawal
Description: Number of Participants with an Adverse Event leading to study drug withdrawal
Time Frame: Test of cure 2 (up to approximately 42 days)
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Algorithm-determined Therapy
Number analyzed (Participants) | 254 | 255
Participants | 1 | 4

4. Primary Outcome: Number of Participants That Changed From Vancomycin to Another Study Antibiotic Due to an Adverse Event
Description: Patient changes from vancomycin or a protocol-approved study antibiotic to another protocol-approved study antibiotic due to AE associated with study drug
Time Frame: Test of cure 2 (up to approximately 42 days)
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Algorithm-determined Therapy
Number analyzed (Participants) | 254 | 255
Participants | 2 | 5

5. Secondary Outcome: Antibiotic Days by Treatment Group
Description: This will be analyzed by evaluating the difference in antibiotic days by treatment group and calculating 95% confidence intervals around the difference in antibiotic days among study patients randomized to algorithm-based treatment vs. among study patients randomized to standard treatment.
Time Frame: Test of cure 2 (up to approximately 42 days)
Population: PP (per protocol) population and PPE Population: Patients from the PP population who did not have complicated staphylococcal infection.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard of Care | Algorithm-determined Therapy
Number analyzed (Participants) | 203 | 207
Days
  PP Population | 7.9 (8.8) | 7.5 (10.0)
  PPE Population: number analyzed (Participants) | 183 | 171
  PPE Population | 6.2 (6.6) | 4.4 (5.5)

ADVERSE EVENTS:
Time Frame: Baseline until the final TOC (test of cure, up to approximately 42 days).
Arm/Group | Standard of Care | Algorithm-determined Therapy
All-Cause Mortality (participants affected / at risk) | 14/254 | 16/255
Serious Adverse Events (participants affected / at risk) | 72/254 | 83/255
Other Adverse Events (participants affected / at risk) | 6/254 | 7/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=254) | Algorithm-determined Therapy (N=255)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 5 (7)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 6 (6) | 4 (4)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 7 (7)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 1 (2) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 9 (9)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=254) | Algorithm-determined Therapy (N=255)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2013-12-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT01191840/SAP_000.pdf
  • Study Protocol: Amendment 4 (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT01191840/Prot_001.pdf
  • Informed Consent Form: Amendment 4 ICF (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT01191840/ICF_002.pdf